CLINICAL TRIAL: NCT02859441
Title: A Phase I/II Trial for Intravitreous Treatment of Severe Ocular Von Hippel-Lindau Disease Using a Combination of the PDGF Antagonist E10030 and the VEGF Antagonist Ranibizumab
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160159; 16-EI-0159
Record Dates: First submitted 2016-08-06; First posted 2016-08-09 (Estimated); Results first posted 2020-07-14 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2019-07

CONDITIONS: Von Hippel-Lindau Syndrome
Keywords: Intravitreal Injection; Retinal Capillary Hemangioma
MeSH Terms: conditions — von Hippel-Lindau Disease | interventions — Ranibizumab; E10030 aptamer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- E10030 and Ranibizumab (Experimental): Intravitreal injections of E10030 and Ranibizumab
  Interventions: Drug: Ranibizumab; Drug: E10030

INTERVENTIONS:
Drug: Ranibizumab — Intravitreal injections of the commercially-available 10 mg/mL formulation of ranibizumab. Ranibizumab is formulated as a sterile solution (pH 5.5) with histidine, trehalose and polysorbate 20. The vial contains no preservative. Each vial contains 0.5 mL of 10 mg/mL ranibizumab aqueous solution. The intravitreal injection volume of ranibizumab is 50 microliter, which correlates to 0.5 mg of dry ranibizumab.
Drug: E10030 — E10030 is not a commercially available drug product, and will be provided by Ophthotech Corp. The drug product is provided as a sterile aqueous solution of E10030 at a concentration of 30 mg (oligo weight)/mL. The solution contains monobasic sodium phosphate monohydrate and dibasic sodium phosphate heptahydrate as buffering agents as well as sodium chloride as a tonicity adjuster. The intravitreal injection volume of E10030 is 50 microliter, which correlates to 1.5 mg of dry E10030.

SUMMARY:
Background: People with Von-Hippel-Lindau (VHL) disease may experience significant vision loss as a result of retinal capillary hemangiomas (RCH), the most common and often earliest manifestation of VHL.

Objective: To investigate the safety and possible efficacy of combination investigational treatment with serial intravitreal injections of E10030, a PDGF-B antagonist, and ranibizumab, a VEGF-A antagonist, in participants with severe ocular VHL disease.

Design: Three participants with severe ocular VHL disease will receive the combination investigational treatment in one eye and will be followed for 104 weeks.

Primary Outcome: The safety of the combination investigational treatment, assessed by tabulation of adverse events reported through Week 52.

DETAILED DESCRIPTION:
Objective: Von Hippel-Lindau (VHL) disease is an autosomal dominant heritable disorder in which multiple benign and malignant neoplasms and cysts of specific histopathologies develop in the kidney, adrenal gland, pancreas, brain, spinal cord, eye, inner ear, epididymis and broad ligament. The disease affects about 7,000 individuals in the United States. Retinal capillary hemangiomas (RCH) are the most common and often the earliest manifestation of VHL disease and may lead to significant vision loss. In some such eyes, inexorable progression of RCH leads to blindness and phthisis bulbi despite aggressive treatment. Levels of vascular endothelial growth factor (VEGF), a potent mediator of angiogenesis and vascular permeability, have been shown to be elevated in multiple cell types deficient in the VHL protein (pVHL). Platelet-derived growth factor (PDGF), which has an important role in stabilization of immature new vessels during angiogenesis, is upregulated in pVHL-defective cell lines and expressed in other pVHL-defective tumors. Anti-VEGF therapy alone had no beneficial effect on ocular VHL disease in two previous phase 1 studies. The objective of this study is to investigate the safety and possible efficacy of combination investigational treatment with serial intravitreal injections of E10030, a PDGF-B antagonist, and ranibizumab, a VEGF-A antagonist, in participants with severe ocular VHL disease.

Study Population: Three participants with severe ocular VHL disease will receive the combination investigational treatment in one eye and will be followed for 104 weeks.

Design: In this phase I/II, single-center, prospective, open label, non-randomized, uncontrolled, single group trial, one eye of eligible participants will be treated with investigational products, E10030, a PDGF-B antagonist, and ranibizumab, a VEGF-A antagonist. Participants will receive combination investigational treatment consisting of intravitreal injections of E10030 (1.5 mg in 0.05 mL) and ranibizumab (0.5 mg in 0.05 mL) every four weeks from baseline through Week 16 (totaling five treatments) and then every eight weeks through Week 48 (totaling nine treatments from baseline). All participants will be followed for 104 weeks.

Outcome Measures: The primary outcome for the study will be safety of the combination investigational treatment, assessed by tabulation of adverse events reported through Week 52. Secondary outcomes will include tabulation of adverse events at Week 104, and the following measures in the study eye at Week 52 and 104: the proportion of participants experiencing reduction in size of at least one RCH in the absence of other ablative treatment (assessed by fundus photography and fluorescein angiography (FA)); the proportion of participants experiencing moderate vision loss (defined as a loss of greater than or equal to 15 letters from baseline on Electronic Visual Acuity (EVA) testing); mean change in visual acuity; change in size of RCH (measured by fundus photography and FA); change in exudation (measured by fundus photography, optical coherence tomography (OCT) and FA); change in epiretinal proliferation, fibrosis or retinal traction (assessed by OCT and fundus photography); proportion of participants undergoing ablative treatment of RCH or ocular surgery; proportion of participants with successful ablative treatment of RCH; and the proportion of participants with appearance of one or more new RCH.

ELIGIBILITY:
* Participant Eligibility Criteria

The participant must meet all of the eligibility criteria and none of the exclusion criteria below.

INCLUSION CRITERIA:

1. Participant must understand and sign the informed consent.
2. Participant must be 18 years of age or older.
3. Participant must have a diagnosis of VHL disease. In accordance with established criteria for diagnosis, any one of the following will be considered sufficient evidence that VHL disease is present:

   * A family history of VHL disease plus one or more of the following lesions: RCH, spinal or cerebellar hemangioblastoma, pheochromocytoma, multiple pancreatic cysts, epididymal or broad ligament cystadenomas, multiple renal cysts or renal cell carcinoma before age 60 years.
   * Presence of two or more hemangioblastomas of the retina or brain or a single hemangioblastoma in association with a visceral manifestation such as kidney or pancreatic cysts; renal cell carcinoma; adrenal or extra-adrenal pheochromocytomas; endolymphatic sac tumors; papillary cystadenomas of the epididymis or broad ligament; or neuroendocrine tumors of the pancreas.
   * Presence of a known disease-causing germline mutation in the VHL gene.
4. Any female participant of childbearing potential must not be pregnant or breast-feeding, must have a negative pregnancy test at screening and must be willing to undergo pregnancy testing immediately prior to each treatment.
5. Any female participant of childbearing potential and any male participant able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two effective methods of contraception throughout the course of the study and for at least two months following the last administration of combination investigational treatment. Acceptable methods of contraception include:

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm or condom) with spermicide, or
   * surgical sterilization (hysterectomy, tubal ligation or vasectomy).

EXCLUSION CRITERIA:

1. Participant has a history or evidence of significant cardiac disease (for example, use of cardiac medications aside from agents to control blood pressure, past acute coronary syndrome, past myocardial infarction, past revascularization procedure or arrhythmias requiring past or present treatment).
2. Participant has a history of stroke or transient ischemic attack.

   Note: cerebrovascular manifestations and/or complications of central nervous system hemangioblastomas are not exclusionary, in the absence of past stroke or transient ischemic attack.
3. Participant has used systemic medication with significant anti-VEGF or anti-PDGF activity within 30 days of study entry or expects use of such a medication within 12 months of study entry.
4. Participant is medically unable to comply with study procedures or follow-up in the judgment of the investigator.
5. Participant has a diagnosis of diabetic mellitus (type 1 or type 2). Any one of the following will be considered sufficient evidence that diabetes is present:

   * Current regular use of insulin for the treatment of diabetes,
   * Current regular use of oral anti-hyperglycemia agents for the treatment of diabetes,
   * Hemoglobin A1C of greater than or equal to 6.5%, or
   * Documented diabetes by the American Diabetes Association (ADA) and/or World Health Organization (WHO) criteria.

Study Eye Eligibility Criteria

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

INCLUSION CRITERIA:

1. Participant has at least one RCH secondary to VHL disease in the study eye that fulfills the following criteria:

   1. The RCH must exhibit growth potential with consequent threat to vision. Growth potential with consequent threat to vision is defined by AT LEAST ONE of the following:

      * Associated intra- or sub-retinal exudation or lipid deposition that, in the judgment of the investigator, reflects ongoing vascular incompetence and is not solely reflective of residual changes following previous treatment or solely secondary to coexistent retinal traction.
      * Increased size of the tumor compared to a previous time point as assessed by fundus photography or FA.
      * Associated intra-, sub- or pre-retinal hemorrhage not secondary to previous treatment, as assessed by fundus photography or FA.
      * The presence of dilated and/or tortuous feeder vessels.
      * Vitreous cell or haze indicative of vitreous exudation, in the absence of other ocular features potentially responsible for such findings.
   2. The RCH, in the judgment of the investigator, is NOT readily treatable using thermal laser because of its size, posterior location, poor previous response to conventional therapy, association with significant exudation, epiretinal proliferation, associated vascular abnormalities such as vascular proliferation or diffusely incompetent retinal vessels, or other factors predictive of a poor response to standard of care approaches.
2. The study eye must have clarity of ocular media and degree of pupil dilation sufficient to permit adequate fundus photography.

EXCLUSION CRITERIA:

1. The study eye has present or chronic ocular or periocular infection (including any history of ocular herpes zoster).
2. The study eye has chronic glaucoma; OR has received anti-glaucoma medication at any time within 90 days of study entry; OR has significant ocular hypertension, defined as documented intraocular pressure of greater than or equal to 28 mmHg on any occasion in the absence of self-limited acute glaucoma, OR greater than or equal to 24 mmHg on at least two occasions in the absence of self-limited acute glaucoma.

   Note: History of self-limited acute glaucoma in a study eye, if now resolved and not expected to recur, is not exclusionary. History of glaucoma or ocular hypertension in the fellow eye, if not felt to significantly impact risk of glaucoma in the study eye, is not exclusionary.
3. The study eye has undergone any surgical procedure within 60 days prior to study entry (inclusive of cryotherapy or thermal laser).
4. The study eye has a history of intravitreal injection of an anti-VEGF agent (such as bevacizumab, ranibizumab or aflibercept) within 42 days prior to study entry.
5. The study eye has a history of intravitreal or periocular injection of long-acting corticosteroids (such as triamcinolone acetonide) within 90 days of study entry or history of any sustained-release ocular drug delivery device with reasonable expectation of residual activity in the study eye.

Choice of Study Eye in Cases of Bilateral Eligibility

If both eyes of a participant meet the criteria described above, the investigator will choose to enroll one eye in consultation with the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry E Wiley, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Result] Hwang CK, Chew EY, Cukras CA, Keenan TDL, Wong WT, Linehan WM, Chittiboina P, Pacak K, Wiley HE. Intravitreous treatment of severe ocular von Hippel-Lindau disease using a combination of the VEGF inhibitor, ranibizumab and PDGF inhibitor, E10030: Results from a phase 1/2 clinical trial. Clin Exp Ophthalmol. 2021 Dec;49(9):1048-1059. doi: 10.1111/ceo.14001. Epub 2021 Oct 26. PMID 34549489
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-EI-0159.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E10030 and Ranibizumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 44.7 [35 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Tabulation of Adverse Events
Description: The total number of adverse events through Week 52.
Time Frame: From Baseline to Week 52
Measure: Number; unit: adverse events
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
adverse events | 13

2. Secondary Outcome: Tabulation of Adverse Events
Description: The total number of adverse events, excluding natural progression of disease events, through Week 104.
Time Frame: From Baseline to Week 104
Measure: Number; unit: adverse events
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
adverse events | 27

3. Secondary Outcome: The Proportion of Participants Experiencing Reduction in Size of at Least One Retinal Capillary Hemangioma (RCH), in the Absence of Other Ablative Treatment (Assessed by Fundus Photography and Fluorescein Angiography (FA))
Description: The proportion of participants experiencing a reduction in size of at least one RCH in the study eye, in the absence of other ablative treatment as assessed by fundus photography and fluorescein angiography (FA), between Baseline and Week 52.
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: The Proportion of Participants Experiencing Reduction in Size of at Least One RCH, in the Absence of Other Ablative Treatment (Assessed by Fundus Photography and Fluorescein Angiography [FA])
Description: The proportion of participants experiencing a reduction in size of at least one RCH in the study eye, in the absence of other ablative treatment as assessed by fundus photography and fluorescein angiography (FA), between Baseline and Week 104.
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Proportion of Participants Undergoing Ablative Treatment of RCH or Ocular Surgery
Description: The proportion of participants undergoing ablative treatment of RCH or ocular surgery in the study eye between Baseline and Week 52.
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

6. Secondary Outcome: Proportion of Participants Undergoing Ablative Treatment of RCH or Ocular Surgery
Description: The proportion of participants undergoing ablative treatment of RCH or ocular surgery in the study eye between Baseline and Week 104.
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

7. Secondary Outcome: Proportion of Participants With Successful Ablative Treatment of RCH
Description: The proportion of participants with successful ablative treatment of RCH in the study eye between Baseline and Week 52.
Time Frame: From Baseline to Week 52
Population: No participants were analyzed for this outcome because none of the participants underwent ablative treatment of RCH. Therefore, no data was collected for this outcome.
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 0

8. Secondary Outcome: Proportion of Participants With Successful Ablative Treatment of RCH
Description: The proportion of participants with successful ablative treatment of RCH in the study eye between Baseline and Week 104.
Time Frame: From Baseline to Week 104
Population: as for outcome 7
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 0

9. Secondary Outcome: Mean Change in Visual Acuity
Description: Mean change in visual acuity in the study eye from Baseline as compared to Week 52 as measured using the Electronic Early Treatment of Diabetic Retinopathy Study (ETDRS) Visual Acuity (EVA) Testing protocol. Acuity is measured as letters read using an electronic ETDRS program.
Time Frame: Baseline and Week 52
Population: Mean visual acuity values are presented for Baseline and Week 52 and the mean change at Week 52 from Baseline for the study eye.
Measure: Mean (Standard Deviation); unit: Letters Read
Groups:
- Visual Acuity at Baseline; Visual Acuity at Week 52; Mean Change in Visual Acuity at Week 52 From Baseline: Intravitreal injections of E10030 and Ranibizumab
Arm/Group | Visual Acuity at Baseline | Visual Acuity at Week 52 | Mean Change in Visual Acuity at Week 52 From Baseline
Number analyzed (Participants) | 3 | 3 | 3
Letters Read | 64.0 (26.3) | 59.0 (21.3) | -5.0 (7.0)

10. Secondary Outcome: Mean Change in Visual Acuity
Description: Mean change in visual acuity in the study eye from Baseline as compared to Week 104 as measured using the Electronic Early Treatment of Diabetic Retinopathy Study (ETDRS) Visual Acuity (EVA) Testing protocol. Acuity is measured as letters read using an electronic ETDRS program.
Time Frame: Baseline and Week 104
Population: Mean visual acuity values are presented for Baseline and Week 104 and the mean change at Week 104 from Baseline for the study eye.
Measure: Mean (Standard Deviation); unit: Letters Read
Groups:
- Visual Acuity at Week 104; Mean Change in Visual Acuity at Week 104 From Baseline: Intravitreal injections of E10030 and Ranibizumab
Arm/Group | Visual Acuity at Baseline | Visual Acuity at Week 104 | Mean Change in Visual Acuity at Week 104 From Baseline
Number analyzed (Participants) | 3 | 3 | 3
Letters Read | 64.0 (26.3) | 45.0 (40.1) | -19.0 (14.1)

11. Secondary Outcome: The Proportion of Participants Experiencing Moderate Vision Loss (Defined as a Loss of Greater Than or Equal to 15 Letters From Baseline on Electronic Visual Acuity [EVA] Testing)
Description: The proportion of participants experiencing moderate vision loss in the study eye (defined as a loss of greater than or equal to 15 letters from baseline on Electronic Visual Acuity [EVA] testing) between Baseline and Week 52.
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

12. Secondary Outcome: The Proportion of Participants Experiencing Moderate Vision Loss (Defined as a Loss of Greater Than or Equal to 15 Letters From Baseline on Electronic Visual Acuity [EVA] Testing)
Description: The proportion of participants experiencing moderate vision loss in the study eye (defined as a loss of greater than or equal to 15 letters from baseline on Electronic Visual Acuity [EVA] testing) between Baseline and Week 104.
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 2

13. Secondary Outcome: Change in Size of RCH (Measured by Fundus Photography and FA)
Description: Number of participants who experienced increased, decreased, or mixed change in the size of RCH in the study eye between Baseline and Week 52 (measured by fundus photography and FA).
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Groups:
- Increase in Size of RCH; Decrease in Size of RCH; Mixed Change in Size of RCH; No Change in Size of RCH: Intravitreal injections of E10030 and Ranibizumab
Arm/Group | Increase in Size of RCH | Decrease in Size of RCH | Mixed Change in Size of RCH | No Change in Size of RCH
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 2

14. Secondary Outcome: Change in Size of RCH (Measured by Fundus Photography and FA)
Description: Number of participants who experienced increased, decreased, or mixed change in the size of RCH in the study eye between Baseline and Week 104 (measured by fundus photography and FA).
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | Increase in Size of RCH | Decrease in Size of RCH | Mixed Change in Size of RCH | No Change in Size of RCH
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 2

15. Secondary Outcome: Change in Exudation (Measured by Fundus Photography, Optical Coherence Tomography (OCT) and FA)
Description: Number of participants who experienced increased, decreased, or mixed change in exudation in the study eye between Baseline and Week 52 (measured by fundus photography, optical coherence tomography [OCT] and FA).
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Groups:
- Increased Exudation; Decreased Exudation; Mixed Change in Exudation; No Change in Exudation: Intravitreal injections of E10030 and Ranibizumab
Arm/Group | Increased Exudation | Decreased Exudation | Mixed Change in Exudation | No Change in Exudation
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 1

16. Secondary Outcome: Change in Exudation (Measured by Fundus Photography, Optical Coherence Tomography [OCT] and FA)
Description: Number of participants who experienced increased, decreased, or mixed change in exudation in the study eye between Baseline and Week 104 (measured by fundus photography, optical coherence tomography [OCT] and FA).
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | Increased Exudation | Decreased Exudation | Mixed Change in Exudation | No Change in Exudation
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 1 | 1

17. Secondary Outcome: Change in Epiretinal Proliferation, Fibrosis or Retinal Traction (Assessed by OCT and Fundus Photography)
Description: Number of participants who experienced increased, decreased, or mixed change in epiretinal proliferation, fibrosis or retinal traction in the study eye between Baseline and Week 52 (assessed by OCT and fundus photography).
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Groups:
- Increased Change; Decreased Change; Mixed Change; No Change: Intravitreal injections of E10030 and Ranibizumab
Arm/Group | Increased Change | Decreased Change | Mixed Change | No Change
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 2

18. Secondary Outcome: Change in Epiretinal Proliferation, Fibrosis or Retinal Traction (Assessed by OCT and Fundus Photography)
Description: Number of participants who experienced increased, decreased, or mixed change in epiretinal proliferation, fibrosis or retinal traction in the study eye between Baseline and Week 104 (assessed by OCT and fundus photography).
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | Increased Change | Decreased Change | Mixed Change | No Change
Number analyzed (Participants) | 3 | 3 | 3 | 3
Participants | 1 | 0 | 0 | 2

19. Secondary Outcome: Proportion of Participants With Appearance of One or More New RCH
Description: The proportion of participants with appearance of one or more new RCH in the study eye between Baseline and Week 52.
Time Frame: From Baseline to Week 52
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 0

20. Secondary Outcome: Proportion of Participants With Appearance of One or More New RCH
Description: The proportion of participants with appearance of one or more new RCH in the study eye between Baseline and Week 104.
Time Frame: From Baseline to Week 104
Measure: Count of Participants; unit: Participants
Arm/Group | E10030 and Ranibizumab
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: 104 Weeks
Description: Adverse events were collected on and after the baseline visit.
Arm/Group | E10030 and Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 and Ranibizumab (N=3)
Nephrolithiasis (Renal and urinary disorders) | 1 (2) — Nephrolithiasis
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Severe Dehydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E10030 and Ranibizumab (N=3)
Ocular Hypertension (Eye disorders) | 1 (3) — Mild Ocular Hypertension
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Lower Back Pain
Hypoaesthesia (Nervous system disorders) | 1 (1) — Left Foot Numbness
Infection (Infections and infestations) | 1 (1) — Infection
Posterior Capsule Opacification (Eye disorders) | 1 (1) — Capsular opacity,OD
Visual Acuity Reduced (Eye disorders) | 2 (3) — Decrease in Visual Acuity
Vomiting (Gastrointestinal disorders) | 1 (1) — Vomiting
Weight Decreased (Investigations) | 1 (1) — Weight Loss
Eye Pain (Eye disorders) | 1 (1) — Periocular Pain/Brow Headache
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) — Right Foot Injury
Vitreous Haemorrhage (Eye disorders) | 1 (1) — Mild Vitreous Haemorrhage
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Upper Respiratory Inflammation
Pyrexia (General disorders) | 1 (1) — Fever
Corneal Abrasion (Eye disorders) | 1 (1) — Corneal Abrasion
Keratopathy (Eye disorders) | 1 (2) — Decreased Vision due to Band Keratopathy
Corneal Erosion (Eye disorders) | 1 (1) — Corneal Erosion
Corneal Neovascularization (Eye disorders) | 1 (1) — Corneal Neovascularization
Blood Pressure Increased (Investigations) | 1 (1) — Elevated Blood Pressure
Retinal Haemorrhage (Eye disorders) | 1 (1) — Dot Intraretinal Haemorrhage
Von Hippel-Lindau Disease (Congenital, familial and genetic disorders) | 1 (1) — Treatment of Von Hippel-Lindau lesions in fellow eye with laser (Natural Progression of Disease Event)
Haemangioma of Retina (Congenital, familial and genetic disorders) | 1 (1) — Small new retinal hemangioma in OD (Natural Progression of Disease Event)
Iris Adhesions (Eye disorders) | 1 (1) — Focal posterior synechiae, left eye (Natural Progression of Disease Event)
Eye Laser Surgery (Surgical and medical procedures) | 1 (1) — Laser of pre-existing Von Hippel-Lindau lesion in fellow eye (Natural Progression of Disease Event)
Eye Haemorrhage (Eye disorders) | 1 (1) — Mild intraocular hemorrhage, right eye (Natural Progression of Disease Event)
Iris Neovascularisation (Eye disorders) | 1 (1) — Iris neovascularization, right eye (Natural Progression of Disease Event)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT02859441/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT02859441/SAP_001.pdf